CLINICAL TRIAL: NCT06620913
Title: Clinico-immunological Characterization and Immune Tolerance Breakdown in CV2-autoimmunity
Acronym: CarTo-CV2
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5225
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: CV2 Autoimmunity
Keywords: Paraneoplastic neurological disorders, lung cancer, CV2 autoimmunity, immune tolerance breakdown
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, PBMCs, DNA, CSF and tumor collected at the time of diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CV2 Abs: Patients harboring CV2 Abs and a paraneoplastic neurological syndromes.
  Interventions: Other: Description of clinical, immunological and tumor features of patients harboring CV2 Abs

INTERVENTIONS:
Other: Description of clinical, immunological and tumor features of patients harboring CV2 Abs — This is a non-interventional study involving clinical data and biological samples (DNA and tumors block). Demographic and clinical data already collected in the database of the French Reference Center on PNS will be reviewed. The diagnostic tests performed to detect CV2-Abs in the patients already included in the database of the French Reference Center on PNS will be retrospectively analyzed.

SUMMARY:
Paraneoplastic neurological syndromes are rare syndromes caused by the remote effects of cancer. They have an immune-mediated pathogenesis, yet the underlying mechanisms are not fully elucidated. CV2/Collapsin response-mediator protein 5 (CRMP5)-IgG paraneoplastic neurological syndrome is characterized by heterogeneous clinical presentations, affecting both central and peripheral nervous system, and the most frequently associate tumor is small cell lung carcinoma. Central nervous system involvement along with CSF and neuroimaging findings have not been fully described in the literature in CV2/CRMP5 patients. Unraveling the complexities of CV2/CRMP5 paraneoplastic neurological syndrome is critical to improve diagnosis, treatment, and patients' care. Our intention is to perform a comprehensive analysis of the clinical characteristics and instrumental investigations of a large cohort of CV2/CRMP5 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with paraneoplastic neurological syndromes
* Patient with CV2 antibody in sera and/or CSF

Exclusion Criteria:

* Patient with no data
* Patient without neurological disorder
* Patient without CV2 antibody in sera/CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients harboring CV2 Abs in serum and/or CSF with or without cancer.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRs) | At baseline, 3, 6, 12, 18 month
  Application of modified rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Pr Jérôme Honnorat, Pr, Principal Investigator — Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France.
Locations (1):
- Hôpital Neurologique Pierre Wertheimer / Groupement Hospitalier Est, Bron, France